CLINICAL TRIAL: NCT03595488
Title: Dupilumab as add-on Therapy for Aspirin-exacerbated Respiratory Disease (AERD)
Brief Title: Dupilumab for Aspirin-exacerbated Respiratory Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rochester General Hospital (Other)
Responsible Party: Principal Investigator, S. Shahzad Mustafa, Principle Investigator, Rochester General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1828-A-18
Record Dates: First submitted 2018-06-29; First posted 2018-07-23 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Aspirin-exacerbated Respiratory Disease
MeSH Terms: interventions — dupilumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Single-blinded, Dupilumab or matching placebo will be administered to the patients at the study visits. At each study visit, a single dose of dupilumab or placebo will be dispensed to the patients to be administered at home.
  300 mg/2 ml solution in a single-dose pre-filled syringe with needle shield given once every 2 weeks in a subcutaneous injection
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — dupilumab 300 mg subcutaneous injection every 2 weeks
  Other Names: Matching placebo

SUMMARY:
Subjects with physician-diagnosed aspirin-exacerbated respiratory disease (AERD) who remain unacceptably symptomatic with a SNOT 22 score > 18 despite routine medical therapy will be enrolled in this single center, single-blinded study assessing the efficacy of dupilumab in AERD.

DETAILED DESCRIPTION:
This is a single blind, placebo controlled trial to be conducted in adult patients with AERD to determine the efficacy and safety of dupilumab in treating symptoms of chronic rhinosinusitis.

All subjects will be treated with the FDA-approved and the commercially available dose for adult atopic dermatitis of 300 mg every 2 weeks administered subcutaneously, based on the observed efficacy and safety of this dose. In addition to atopic dermatitis, this dose has also been shown to be efficacious in adult asthma.15 Patients will not be treated with a loading dose since other studies of dupilumab in asthma and chronic rhinosinusitis with nasal polyposis have not used a loading dose.

There will be a one month screening period to determine the patient's eligibility and establish symptom control and baseline parameters.

Patients will continue their background medications for chronic rhinosinusitis with nasal polyposis and asthma. These medications may include nasal corticosteroids, nasal antihistamines, systemic antihistamines, leukotriene receptor antagonists, 5 lipo-oxygenase inhibitors, inhaled corticosteroids, long-acting beta agonists, and long acting muscarinic antagonists. These controller medications will not be dispensed or supplied by the sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years and older with a physician diagnosis of aspirin-exacerbated respiratory disease, as defined by a physician diagnosis of asthma, chronic rhinosinusitis with nasal polyposis, and a convincing clinical history of NSAID sensitivity
2. All subjects must have a SNOT 22 score ≥ 19 despite standard medical therapy. This minimal SNOT 22 was calculated by taking the range of SNOT 22 scores in studies of normal controls plus 8.9, which is the minimal clinically meaningful improvement in SNOT 22 score detected by patients.
3. Able to understand and willingness to sign informed consent
4. Able to comply with study procedures

Exclusion Criteria:

1. Patient < 18 years of age
2. Pregnancy or breast feeding
3. Current tobacco use
4. Significant, uncontrolled medical conditions
5. Ongoing malignancy or history of malignancy in remission within the past 12 months
6. Current treatment with immunosuppressive medications except chronic oral steroids
7. Currently increasing dose of aeroallergen immunotherapy (patients on stable dose of aeroallergen immunotherapy will be allowed to participate)
8. Treatment with omalizumab, reslizumab, mepolizumab within 4 months of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
SNOT 22 Score | From baseline to completion of study(7 months total)
  This is a patient-reported outcome score for chronic rhinosinusitis with or without nasal polyposis

SECONDARY OUTCOMES:
UPSIT | From baseline to completion of study( 7 months total)
  Univ. of Pennsylvania smell identification test
Lund Mackay score | From baseline to completion of study( 7 months total)
  Objective score for CT sinus imaging, this is a widely used method for radiologic staging of chronic rhinosinusitis.
ACT score | From baseline to completion of study( 7 months total)
  Validated asthma control test, a series of 5 questions related to patient's asthma control over the previous 4 weeks.
Asthma Mini-AQLQ, 15 questions to assess quality of life. This assessment takes approximately 4-5 minutes to complete the questions. | From baseline to completion of study( 7 months total)
  Validated asthma quality of life score
Change in FEV1 | From baseline to completion of study( 7 months total)
  Forced expiratory volume in first second from spirometry
Change in FeNO | From baseline to completion of study( 7 months total)
  Exhaled nitric oxide
Eosinophil count | From baseline to completion of study( 7 months total)
  Absolute eosinophil count
Total serum IgE | From baseline to completion of study( 7 months total)
  Total IgE
Serum tryptase | From baseline to completion of study( 7 months total)
  Biomarker
Serum TARC (thymus and activation regulated cytokine) | From baseline to completion of study( 7 months total)
  Biomarker
Serum prostaglandin D2 | From baseline to completion of study( 7 months total)
  Biomarker
24 hour urinary leukotriene E4 | From baseline to completion of study( 7 months total)
  Biomarker
To assess the safety and tolerability of dupilumab | From baseline to completion of study( 7 months total)
  Adverse events
To assess cumulative dose of systemic steroids | From baseline to completion of study( 7 months total)
  Impact on systemic steroids

CONTACTS AND LOCATIONS:
Overall Officials: S Shahzad Mustafa, MD, Principal Investigator — Lead Physician
Locations (1):
- Rochester Regional Health - Allergy/Immunology, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rajan JP, Wineinger NE, Stevenson DD, White AA. Prevalence of aspirin-exacerbated respiratory disease among asthmatic patients: A meta-analysis of the literature. J Allergy Clin Immunol. 2015 Mar;135(3):676-81.e1. doi: 10.1016/j.jaci.2014.08.020. Epub 2014 Oct 3. PMID 25282015
- [Background] Mullol J, Picado C. Rhinosinusitis and nasal polyps in aspirin-exacerbated respiratory disease. Immunol Allergy Clin North Am. 2013 May;33(2):163-76. doi: 10.1016/j.iac.2012.11.002. Epub 2012 Dec 23. PMID 23639706
- [Background] Ta V, White AA. Survey-Defined Patient Experiences With Aspirin-Exacerbated Respiratory Disease. J Allergy Clin Immunol Pract. 2015 Sep-Oct;3(5):711-8. doi: 10.1016/j.jaip.2015.03.001. Epub 2015 Apr 7. PMID 25858054
- [Background] Berges-Gimeno MP, Simon RA, Stevenson DD. Long-term treatment with aspirin desensitization in asthmatic patients with aspirin-exacerbated respiratory disease. J Allergy Clin Immunol. 2003 Jan;111(1):180-6. doi: 10.1067/mai.2003.7. PMID 12532116
- [Background] Stevenson DD, Pleskow WW, Simon RA, Mathison DA, Lumry WR, Schatz M, Zeiger RS. Aspirin-sensitive rhinosinusitis asthma: a double-blind crossover study of treatment with aspirin. J Allergy Clin Immunol. 1984 Apr;73(4):500-7. doi: 10.1016/0091-6749(84)90361-0. PMID 6368649
- [Background] Swierczynska-Krepa M, Sanak M, Bochenek G, Strek P, Cmiel A, Gielicz A, Plutecka H, Szczeklik A, Nizankowska-Mogilnicka E. Aspirin desensitization in patients with aspirin-induced and aspirin-tolerant asthma: a double-blind study. J Allergy Clin Immunol. 2014 Oct;134(4):883-90. doi: 10.1016/j.jaci.2014.02.041. Epub 2014 Apr 24. PMID 24767875
- [Background] Fruth K, Pogorzelski B, Schmidtmann I, Springer J, Fennan N, Fraessdorf N, Boessert A, Schaefer D, Gosepath J, Mann WJ. Low-dose aspirin desensitization in individuals with aspirin-exacerbated respiratory disease. Allergy. 2013;68(5):659-65. doi: 10.1111/all.12131. Epub 2013 Mar 7. PMID 23464577
- [Background] Esmaeilzadeh H, Nabavi M, Aryan Z, Arshi S, Bemanian MH, Fallahpour M, Mortazavi N. Aspirin desensitization for patients with aspirin-exacerbated respiratory disease: A randomized double-blind placebo-controlled trial. Clin Immunol. 2015 Oct;160(2):349-57. doi: 10.1016/j.clim.2015.05.012. Epub 2015 Jun 14. PMID 26083948
- [Background] Waldram JD, White AA. A survey of aspirin desensitization practices among allergists and fellows in training in the United States. J Allergy Clin Immunol Pract. 2016 Nov-Dec;4(6):1253-1255. doi: 10.1016/j.jaip.2016.06.016. Epub 2016 Jul 21. No abstract available. PMID 27452889
- [Background] Samuelsson B, Dahlen SE, Lindgren JA, Rouzer CA, Serhan CN. Leukotrienes and lipoxins: structures, biosynthesis, and biological effects. Science. 1987 Sep 4;237(4819):1171-6. doi: 10.1126/science.2820055.
- [Background] Laidlaw TM, Boyce JA. Aspirin-Exacerbated Respiratory Disease--New Prime Suspects. N Engl J Med. 2016 Feb 4;374(5):484-8. doi: 10.1056/NEJMcibr1514013. No abstract available. PMID 26840139
- [Background] Bachert C, Zhang N. Chronic rhinosinusitis and asthma: novel understanding of the role of IgE 'above atopy'. J Intern Med. 2012 Aug;272(2):133-43. doi: 10.1111/j.1365-2796.2012.02559.x. PMID 22640264
- [Background] Patou J, Gevaert P, Van Zele T, Holtappels G, van Cauwenberge P, Bachert C. Staphylococcus aureus enterotoxin B, protein A, and lipoteichoic acid stimulations in nasal polyps. J Allergy Clin Immunol. 2008 Jan;121(1):110-5. doi: 10.1016/j.jaci.2007.08.059. Epub 2007 Nov 5. PMID 17980412
- [Background] Wenzel S, Ford L, Pearlman D, Spector S, Sher L, Skobieranda F, Wang L, Kirkesseli S, Rocklin R, Bock B, Hamilton J, Ming JE, Radin A, Stahl N, Yancopoulos GD, Graham N, Pirozzi G. Dupilumab in persistent asthma with elevated eosinophil levels. N Engl J Med. 2013 Jun 27;368(26):2455-66. doi: 10.1056/NEJMoa1304048. Epub 2013 May 21. PMID 23688323
- [Background] Wenzel S, Castro M, Corren J, Maspero J, Wang L, Zhang B, Pirozzi G, Sutherland ER, Evans RR, Joish VN, Eckert L, Graham NM, Stahl N, Yancopoulos GD, Louis-Tisserand M, Teper A. Dupilumab efficacy and safety in adults with uncontrolled persistent asthma despite use of medium-to-high-dose inhaled corticosteroids plus a long-acting beta2 agonist: a randomised double-blind placebo-controlled pivotal phase 2b dose-ranging trial. Lancet. 2016 Jul 2;388(10039):31-44. doi: 10.1016/S0140-6736(16)30307-5. Epub 2016 Apr 27. PMID 27130691
- [Background] Hopkins C, Gillett S, Slack R, Lund VJ, Browne JP. Psychometric validity of the 22-item Sinonasal Outcome Test. Clin Otolaryngol. 2009 Oct;34(5):447-54. doi: 10.1111/j.1749-4486.2009.01995.x. PMID 19793277
- [Background] Doty RL, Shaman P, Dann M. Development of the University of Pennsylvania Smell Identification Test: a standardized microencapsulated test of olfactory function. Physiol Behav. 1984 Mar;32(3):489-502. doi: 10.1016/0031-9384(84)90269-5. PMID 6463130
- [Background] Lund VJ, Kennedy DW. Staging for rhinosinusitis. Otolaryngol Head Neck Surg. 1997 Sep;117(3 Pt 2):S35-40. doi: 10.1016/S0194-59989770005-6. PMID 9334786
- [Background] Nathan RA, Sorkness CA, Kosinski M, Schatz M, Li JT, Marcus P, Murray JJ, Pendergraft TB. Development of the asthma control test: a survey for assessing asthma control. J Allergy Clin Immunol. 2004 Jan;113(1):59-65. doi: 10.1016/j.jaci.2003.09.008. PMID 14713908
- [Background] Juniper EF, Buist AS, Cox FM, Ferrie PJ, King DR. Validation of a standardized version of the Asthma Quality of Life Questionnaire. Chest. 1999 May;115(5):1265-70. doi: 10.1378/chest.115.5.1265. PMID 10334138
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Gillett S, Hopkins C, Slack R, Browne JP. A pilot study of the SNOT 22 score in adults with no sinonasal disease. Clin Otolaryngol. 2009 Oct;34(5):467-9. doi: 10.1111/j.1749-4486.2009.01975.x. PMID 19793280
- [Background] Lange B, Thilsing T, Baelum J, Kjeldsen AD. The Sinonasal Outcome Test 22 score in persons without chronic rhinosinusitis. Clin Otolaryngol. 2016 Apr;41(2):127-30. doi: 10.1111/coa.12481. Epub 2016 Feb 4. PMID 26095903
- [Background] Sommer DD, Hoffbauer S, Au M, Sowerby LJ, Gupta MK, Nayan S. Treatment of aspirin exacerbated respiratory disease with a low salicylate diet: a pilot crossover study. Otolaryngol Head Neck Surg. 2015 Jan;152(1):42-7. doi: 10.1177/0194599814555836. Epub 2014 Oct 24. PMID 25344589
- [Background] Sommer DD, Rotenberg BW, Sowerby LJ, Lee JM, Janjua A, Witterick IJ, Monteiro E, Gupta MK, Au M, Nayan S. A novel treatment adjunct for aspirin exacerbated respiratory disease: the low-salicylate diet: a multicenter randomized control crossover trial. Int Forum Allergy Rhinol. 2016 Apr;6(4):385-91. doi: 10.1002/alr.21678. Epub 2016 Jan 11. PMID 26751262
- [Background] Cho KS, Soudry E, Psaltis AJ, Nadeau KC, McGhee SA, Nayak JV, Hwang PH. Long-term sinonasal outcomes of aspirin desensitization in aspirin exacerbated respiratory disease. Otolaryngol Head Neck Surg. 2014 Oct;151(4):575-81. doi: 10.1177/0194599814545750. Epub 2014 Aug 12. PMID 25118195
- [Background] Bachert C, Mannent L, Naclerio RM, Mullol J, Ferguson BJ, Gevaert P, Hellings P, Jiao L, Wang L, Evans RR, Pirozzi G, Graham NM, Swanson B, Hamilton JD, Radin A, Gandhi NA, Stahl N, Yancopoulos GD, Sutherland ER. Effect of Subcutaneous Dupilumab on Nasal Polyp Burden in Patients With Chronic Sinusitis and Nasal Polyposis: A Randomized Clinical Trial. JAMA. 2016 Feb 2;315(5):469-79. doi: 10.1001/jama.2015.19330. PMID 26836729